CLINICAL TRIAL: NCT01749800
Title: Combining Galvanic Vestibular Stimulation and Motor Training in Traumatic Brain Injury Survivors With Attentional Deficits
Brief Title: Galvanic Vestibular Stimulation and Motor Training in Traumatic Brain Injury Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Lab, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-P-000010
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: TBI; Attention Deficits; Motor Impairments
Keywords: TBI; Attention deficits; Upper extremity weakness
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive test with/without GVS (Experimental): Subjects with attention span deficits and no significant motor impairments undergo solely a cognitive test. The test is carried out in multiple trials. For some of the trials (randomly selected), subjects receive galvanic vestibular stimulation (GVS). For other trials, subjects received sham GVS. GVS is delivered using a device by A-M Systems.
  Interventions: Device: GVS; Device: Sham GVS
- Armeo Spring +GVS (Active Comparator): Subjects with both attention span deficits and significant motor impairments undergo robot-assisted upper-limb rehabilitation in combination with galvanic vestibular stimulation (GVS). Robot-assisted training is carried out using the Armeo Spring system by Hocoma AG. GVS is delivered using a device by A-M Systems.
  Interventions: Device: GVS; Device: Armeo Spring
- Armeo Spring + sham GVS (Sham Comparator): Subjects with both attention span deficits and significant motor impairments undergo robot-assisted upper-limb rehabilitation in combination with sham GVS. Robot-assisted training is carried out using the Armeo Spring system by Hocoma AG. Sham stimulation is delivered by connecting the subject to a device by A-M Systems, but the device is not active.
  Interventions: Device: Sham GVS; Device: Armeo Spring

INTERVENTIONS:
Device: GVS — A small current is delivered to the vestibular system via electrodes placed over the subject's mastoid processes.
  Other Names: Device: Model 2200 Analog Stimulus Isolator; Produce by: A-M Systems, Inc., WA, USA
  Arms: Armeo Spring +GVS; Cognitive test with/without GVS
Device: Sham GVS — Electrodes are placed over the subject's mastoid processes and connected to the device, but the device is not active.
  Other Names: Device: Model 2200 Analog Stimulus Isolator; Produce by: A-M Systems, Inc., WA, USA
  Arms: Armeo Spring + sham GVS; Cognitive test with/without GVS
Device: Armeo Spring — A robotic system supports the weak arm of the subject to make it easier to perform therapeutic exercises.
  Other Names: Device: Armeo Spring; Produced by: Hocoma
  Arms: Armeo Spring + sham GVS; Armeo Spring +GVS

SUMMARY:
The overall goal of the proposed project is to perform a preliminary study to assess the potential effects of galvanic vestibular stimulation (GVS) on the outcomes of a cognitive test of attention and the outcomes of robot-assisted upper-limb rehabilitation.

DETAILED DESCRIPTION:
We plan to explore the use of GVS on the severity of attention span deficits and motor training delivered using a spring-based robot. We intend to carry out the study in a small cohort of traumatic brain injury (TBI) survivors (20 subjects). Subjects with attention span deficits but no significant motor impairments will solely undergo a cognitive test of attention with/without GVS. Subjects with both attention span deficits and significant motor impairments will undergo a cognitive test of attention and robot-assisted upper-limb rehabilitation with/without GVS.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe traumatic brain injury involving cognitive and/or motor deficits.
* Neurological injury >1 year prior to study enrollment
* Significant attention deficit
* For subjects with motor deficits (arms 2 and 3), sufficient voluntary movement and range of motion in the most-affected upper extremity to use the robotic arm system (Armeo Spring)

Exclusion Criteria:

* Pregnancy
* History of seizures within 6 months of study enrollment
* Major depression
* Cognitive impairment that may interfere with understanding instructions
* Severe limitations of upper extremity range of motion
* Agitation
* Other major neurological or psychiatric diseases
* Participation in other forms of therapy/ intervention for upper extremity motor recovery
* End-stage liver, kidney, cardiac or pulmonary disease
* A terminal medical diagnosis with survival <1 year
* History of drug or alcohol abuse in the last 3 years
* Adjustment of, or plan to adjust, psychoactive medications within the preceding 1 month, or within the study period.
* Current participation in another interventional trial targeting TBI
* Previous GVS treatment
* Contraindications to GVS such as implants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Test With/Without GVS | Armeo Spring +GVS | Armeo Spring + Sham GVS
Started | 6 (3 subjects did not show significant attention span deficit (required inclusion criterion)) | 1 (1 subject showed significant motor impairments but decided to undergo therapy (exclusion criterion)) | 0
Completed | 3 | 0 | 0
Not Completed | 3 | 1 | 0
Not completed — not meeting inclusion criteria | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Test With/Without GVS | Armeo Spring +GVS | Armeo Spring + Sham GVS | Total
Number analyzed (Participants) | 6 | 1 | 0 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 0 | 7
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 6 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 1 | 0 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 |  | 7
Sustained Attention to Response Task [Mean (Full Range); unit: percentage error] — Subjects are presented with objects (one at the time) on a computer screen and are instructed to press a key on the keyboard according to the characteristics of the object shown on the computer screen. Error rates are measured as percentage of erroneous key selections.
  percentage error | 23 [7 to 33] | 20 [20 to 20] |  | 22 [7 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Sustained Attention to Response Task
Description: Subjects are presented with objects (one at the time) on a computer screen and are instructed to press a key on the keyboard according to the characteristics of the object shown on the computer screen. Error rates are measured as percentage of erroneous key selections.
Time Frame: Baseline and end-of-treatment data (up to 2 weeks)
Measure: Mean (Full Range); unit: percentage errors
Arm/Group | Cognitive Test With/Without GVS | Armeo Spring +GVS | Armeo Spring + Sham GVS
Number analyzed (Participants) | 3 | 0 | 0
percentage errors | 26 [7 to 45] |  |

ADVERSE EVENTS:
Time Frame: Data was collected through study completion (i.e. up to two weeks)
Arm/Group | Cognitive Test With/Without GVS | Armeo Spring +GVS | Armeo Spring + Sham GVS
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Test With/Without GVS (N=6) | Armeo Spring +GVS (N=1) | Armeo Spring + Sham GVS (N=0)
Skin damage caused on the stimulation electrodes (General disorders) | 0 (0) | 0 (0) | 0 (0) — Delivering a small current through the skin could cause skin damage in the areas covered by the stimulation electrodes. We inspected the skin under the electrodes multiple times during the experiments to monitor the skin status.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Test With/Without GVS (N=0) | Armeo Spring +GVS (N=1) | Armeo Spring + Sham GVS (N=0)
Skin irritation caused by the straps of the robot (General disorders) | 0 (0) | 0 (0) | 0 (0) — The robotic system used to facilitate motor training is equipped with straps that are attached to the arm of the subject. The straps could cause skin irritation. The "cognitive test" group did not use the robotic system. Thus, no subject was at risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No